CLINICAL TRIAL: NCT00914225
Title: Effect of Long-lasting Insecticide-treated Bednets and a Point-of-use Water Purification Device on HIV Disease Progression Among ART naïve Patients in Kenya
Brief Title: Effect of Bednets and a Water Purification Device on HIV Disease Progression Among ART naïve Patients in Kenya
Acronym: ITN
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Judd Walson, Associate Professor, Global Health, Medicine (Infectious Disease), University of Washington
Other Study IDs: 35464-B; SSC#1554
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infections; Human Immunodeficiency Virus; Malaria; Plasmodium Falciparum; Diarrhea
Keywords: Human immunodeficiency virus; malaria; plasmodium falciparum; diarrhea; helminth; HIV; Treatment naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Malaria; Malaria, Falciparum; Diarrhea | interventions — Water Purification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma HIV RNA Plasma for Malaria PCR
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention: Cohort 1 is the intervention group who received long-lasting insecticide treated bednets and a water filtration device
  Interventions: Other: Bednets and Water Purification
- Comparison: Cohort 2 is the comparison group included from the control arm of the study, "Empiric therapy of helminth coinfection to reduce HIV-1 disease progression" ClinicalTrials.gov identifier: NCT00507221
  As part of the RCT (NCT00507221), we have enrolled 948 HIV infected ART naïve individuals to compare HIV disease progression in those receiving standard of care versus empiric deworming. Subjects are followed for 24 months and have serial measurements of HIV disease progression, and are evaluated serially for evidence of malaria, diarrhea and other co-morbidities. Participants in this study will have been consented for the collection of data on the frequency of malaria and diarrheal disease, their use of a bednet and water filtration and their compliance with TMP/SMX.

INTERVENTIONS:
Other: Bednets and Water Purification — Individuals in the intervention cohort will be provided with a LLIN and water filtration device. Subjects are followed for 24 months and have serial measurements of HIV disease progression. Data are collected every 3 months on the frequency of malaria, diarrhea and other co-morbidities, as well as compliance with LLIN and water filter use.
  Groups: Intervention

SUMMARY:
In many areas of the world most severely affected by the HIV/AIDS pandemic, insect and water-borne diseases such as malaria and diarrheal disease are common causes of illness and death. In addition, diarrhea and malaria are more common and more severe among adults and children infected with HIV. These infections may modulate the immune system, affect the replication of the HIV virus and could result in more rapid HIV disease progression in co-infected individuals. Access to practical, inexpensive and easy to use interventions to prevent these diseases may be effective in delaying HIV progression.

Current Kenya government and World Health Organization guidelines recommend the use of cotrimoxazole (trimethoprim-sulfamethoxazole [TMP/SMX]) to prevent co-infections, including malaria. Despite the provision of TMP/SMX to HIV-infected adults, infections with malaria and pathogens causing diarrhea remain common causes of morbidity and mortality in many resource-limited settings. In addition, TMP/SMX may not prevent all infections with malaria or other pathogens due to alternative mechanisms of action, antimicrobial resistance and non-compliance due to adverse events or other reasons.

We propose a study to evaluate the impact of providing insecticide treated bednets and a simple water filtration device on markers of HIV disease progression among a cohort of ART naïve, HIV infected adults prescribed TMP/SMX in Kenya. In addition, we propose to evaluate the effect of these interventions on malaria and diarrheal disease incidence and on compliance with TMP/SMX.

DETAILED DESCRIPTION:
Introduction and Background:

Among the estimated 22.5 million HIV infected individuals in sub-Saharan Africa, malaria and diarrheal disease are important causes of morbidity and mortality[1]. Preventive care packages that protect against these co-infections may result in decreased HIV associated morbidity and may also delay HIV disease progression[2]. Long lasting insecticidal nets (LLIN) and water purification systems may be practical and effective interventions for reducing malaria and diarrheal disease incidence and delaying disease progression in HIV infected individuals.

The World Health Organization currently recommends TMP/SMX prophylaxis for immunocompromised HIV infected individuals[3]. TMP/SMX is active against a number of pathogens that cause morbidity and mortality amongst HIV infected individuals, including malaria and infectious causes of diarrhea[4]. Randomized clinical trials in HIV infected children and adults demonstrate marked survival benefits with use of TMP/SMX and cotrimoxazole prophylaxis is recommended for people with HIV in the Kenya Ministry of Health guidelines[5]. In addition, observational studies have suggested benefit on markers of HIV disease progression[5, 6].

HIV infected individuals are at increased risk for malaria infection[7]. LLIN have been associated with a 17% reduction in mortality and a 50% reduction in uncomplicated malaria in areas of stable malaria transmission in HIV-uninfected adults and are a cost-effective method of malaria prevention[8, 9]. In HIV infected individuals, TMP/SMX prophylaxis has been shown to decrease episodes of malaria from ~50/100 person-years (p-yrs) to 9 episodes/100 p-yrs[10]. LLIN may provide additive benefit when combined with TMP/SMX in HIV infected individuals. Amongst HIV infected individuals receiving HAART and TMP/SMX, the addition of LLIN resulted in a 42-60% reduction in the incidence of symptomatic malaria[10]. In HIV infected children receiving TMP/SMX, LLIN were associated with marked decreases in malarial parasitemia[11]. LLIN are simple to administer, requiring a single encounter for long term provision of the intervention, and, in contrast to TMP/SMX, do not pose risk to the individuals of drug toxicity or development of resistant microbial flora.

In addition to malaria, diarrheal disease remains a major cause of morbidity and mortality amongst HIV infected individuals in many parts of sub-Saharan Africa[12, 13]. Limited access to clean water for drinking and food preparation results in exposure to numerous bacterial, viral and parasitic agents of diarrheal disease. Prophylaxis with TMP/SMX has been shown to reduce diarrheal episodes in HIV infected adults from 204 to 148 per 100 person-years[6]. Among HIV-infected adults, the provision of purified drinking water resulted in a 25% reduction in the rate of diarrhea per person year. The addition of TMP-SMX in this cohort resulted in a 67% reduction in diarrheal episodes, suggesting an additive benefit of clean water and TMP/SMX in reducing diarrheal incidence among HIV infected individuals[14]. Similar to LLIN, water filtration devices provide benefit by preventing host ingestion of pathogens and are free of concerns regarding drug resistance or toxicity. Water filtration devices may require more intensive use/training/compliance than LLIN and compliance with daily use of these devices may reduce effectiveness.

It is important to determine if the provision of LLIN and a simple microbiological water purification system are able to slow HIV progression and to reduce the incidence of malaria and diarrheal disease when given in combination with TMP/SMX. If beneficial, this combination of interventions may represent a potentially inexpensive and practical intervention to include as part of an optimized prevention package for HIV-infected individuals in Africa.

Justification of the Study:

Antiretroviral therapy (ART) has dramatically improved the lives of millions of individuals. However, many HIV infected individuals do not yet meet criteria for ART initiation or have limited access to HIV care and treatment. In addition, ART is expensive, can be difficult to tolerate and can lead to the development of resistant virus. Identifying inexpensive, practical and safe interventions to delay disease progression may allow HIV infected individuals to remain healthy for longer periods before requiring ART and may reduce morbidity and mortality due to co-infections. To our knowledge, our study will be the first to look at the effects of non-pharmacological interventions to prevent infectious diseases specifically as a means of delaying HIV disease progression in resource limited settings.

Procedures:

Adult men and women participating in or referred to the HIV Care and Treatment Clinics at each of the included sites will be offered eligibility screening. HIV seropositive individuals with a documented CD4 count ≥350 cells/mm3 will be considered potentially eligible. Those who agree to participate, are willing and able to provide informed consent, are WHO stage I or II based on clinical exam and history (or Stage III based on pulmonary TB only and have completed 2 months of first-line TB therapy), are 18 years of age or older and who are not pregnant (based on urine beta-HCG testing if female) will be offered to participate in this study. Pregnancy testing will be performed at each study visit (every three months) for all premenopausal women. Women who become pregnant during the course of the study will continue to be followed.

All invited participants will be required to sign written informed consent prior to enrollment. At enrollment, all participants will complete a standardized questionnaire assessing medical and social history and will undergo a complete physical examination. Blood specimens will be collected for full blood count with differential, malaria diagnostics, TMP/SMX drug levels, measurement of absolute CD4 count and HIV RNA levels.

A detailed questionnaire will also be administered in order to assess socio-economic status, living conditions, level of education completed, sexual behavior and occupation. This questionnaire will also document potential exposures to infectious diseases such as water supply, sanitation facilities, exposure to mosquitoes and use of LLIN. In addition, a detailed clinical history will also be collected to document any prior illnesses or treatments relevant to HIV or co-infections.

Detailed information regarding the location of each participant's current residence and any additional residences that they consider as a primary dwelling will also be collected by field workers at each site. Global positioning system (GPS) coordinates may be collected at the location of each participant's site of primary residence to facilitate patient tracing. This information will be stored as well as any other potential contact information available (such as cell phone numbers) in order that participants may be traced for the purposes of the study.

All enrolled participants will have scheduled three monthly study visits (enrollment, months 3, 6, 9, 12, 15, 18, 21 and 24) at the clinic from which they were enrolled. At each follow up visit, a standardized questionnaire designed to assess any change in socio-demographic variables or clinical history will be performed. A physical examination will also be performed at each visit. Blood will be collected at all visits for determination of asymptomatic malaria infection as well as markers of other infectious and non-infectious disease markers. At the month 6, 12, 18 and 24 visit, blood will also be collected for measurement of full blood count with differential and CD4 count. Measurement of HIV RNA will be collected at enrolment, the 12 month visit and the 24 month visit. All blood will be separated into plasma and PBMC's (peripheral blood mononuclear cells) and stored for future studies. Any future study utilizing stored specimens will obtain approval from both the Kenya Medical Research Institute and the University of Washington Ethical Review Boards.

Individuals who have evidence of clinical malaria and are parasitemic will be treated following standard Kenyan treatment guidelines. Treatment will be provided by study funds at the clinic according to Kenyan standard of care. Asymptomatic patients will be instructed to return to the clinic immediately if fever develops for repeat testing. Study participants will also be encouraged to come to the study clinic when they are sick in between scheduled visits. During these unscheduled visits for illness, participants with clinical features of malaria will undergo rapid diagnostic testing to confirm malaria infection. Participants who are confirmed to have clinical malaria by rapid diagnostic testing will be referred for free treatment as recommended by the Kenya Ministry of Health. In addition, blood will be drawn for PCR, and malaria thick and thin smears at all unscheduled visits for fever.

Each participant will be visited at their declared residence at two randomly determined time points per year during the course of the study period. All participants will be consented for these visits. Participants may consent for participation without consenting for these visits. Participants who do not consent for these visits will not undergo random home visitation. For participants who consent to the random visitations, the field worker visiting the participant will collect information related to the use of the bednet and water filtration device in order to assess compliance. Information on household members recent illness of malaria and diarrhea will be obtained at these visits.

During the course of the 24 month follow up period, some individuals are expected to meet criteria to initiate ART based on CD4 count or clinical staging. All individuals who are enrolled in the study and who initiate ART will provide detailed information regarding their use of ART, adherence and tolerability. This will aid in the clinical management of these individuals and will provide additional data regarding the response to ART in the groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age.
* Participants must not be or have ever been on highly active antiretroviral therapy CD4 count at enrollment of ≥350 cells/mm3
* WHO Stage I or II or Stage III based on pulmonary TB only and have completed 2 months of first-line therapy.
* Participants must be able and willing to participate and give written informed consent
* Participants must be able and willing to return for the scheduled follow-up visits

Exclusion Criteria:

* Age less than 18 years
* CD4 count <350 cells/mm3
* WHO Stage III or IV HIV Disease study (unless stage III for TB and have completed 2 months of first-line therapy)
* Participants must not be pregnant at the time of enrollment (by urine HCG testing)
* Patients with active tuberculosis who are on second or third line therapy or have not completed at least 2 months of first line TB therapy (Participants who have completed two months of first line TB therapy will be eligible for enrolment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will compare markers of HIV disease progression among ART naive individuals receiving LLIN and a simple microbiological water purification system to the control arm of the randomized controlled trial being conducted at the same clinic settings (NCT00507221).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine the effect of LLIN and a simple microbiological water purification system on markers of HIV progression (time to HAART eligibility and changes in CD4 counts) among antiretroviral naïve, HIV infected adults in Kenya. | Mass screening and enrollment in July 2009, followed by two years of follow-up, and up to a year of data analysis.
  PRIMARY AIM (Aim 1): To determine the effect of the intervention, we will evaluate the effect of the provision of LLIN and water filters on markers of disease progression at 12 months. We will compare the time to eligibility for ART between the groups and the time to CD4 counts of less than 200 and 350 respectively using Cox regression analysis models. In addition, we will compare differences between the mean change in CD4 counts at month 12 of follow-up using ANCOVA controlling for baseline CD4 values.

SECONDARY OUTCOMES:
To determine the effect of LLIN and a simple microbiological water purification system on the incidence of malaria and reported diarrheal disease when added to the standard regimen of TMP/SMX among antiretroviral naïve, HIV infected adults in Kenya. | Same as primary outcome.
  Aim 2: To determine the effect of the intervention on the incidence of diarrheal disease and malaria parasitemia, we will compare the frequency of reported diarrheal illness and documented parasitemia between the intervention and comparison groups using poisson regression or generalized estimating equation model.
To determine the durability of provision of an LLIN and a simple microbiological water purification system on markers of disease progression up to 24 months among antiretroviral naïve, HIV infected adults in Kenya. | Same as primary outcome
  Aim 3: To determine the durability of the intervention, we will evaluate the effect of the provision of LLIN and water filters on markers of disease progression up to 24 months. We will compare the time to eligibility for ART between the groups and the time to CD4 counts of less than 200 and 350 respectively using Cox regression analysis models. In addition, we will compare changes in mean CD4 counts overtime between the groups using linear mixed effects models controlling for baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Judd T Walson, MD MPH, Principal Investigator — University of Washington; Benson Singa, MBChB MPH, Principal Investigator — Kenya Medical Research Institute
Locations (2):
- Kenya (2):
  - Kisii Provincial Hospital, Kisii
  - Kisumu District Hospital, UW/KEMRI Research Clinic, Kisumu